CLINICAL TRIAL: NCT07087886
Title: Combined Intervention of Long-term Letter Mentoring and Centralized Summer Camp by University Student Volunteers for Disadvantaged Children: A Randomized Controlled Trial
Acronym: LWCSC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoxuan Liu (Other)
Responsible Party: Sponsor-Investigator, Xiaoxuan Liu, Phd candidate, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZGL202506-9
Record Dates: First submitted 2025-07-16; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Resilience, Psychological
Keywords: Psychological resilience; Disadvantaged adolescents; Letter-writing support; Summer camp intervention; University student volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A two-phase intervention consisting of (1) a 5-day resilience training summer camp and (2) 10-month letter-writing support by university student volunteers.
  Interventions: Behavioral: Combined Resilience Intervention
- Control Group (No Intervention): Participants will not receive the full intervention but will be offered a condensed version after the study ends for ethical consideration.

INTERVENTIONS:
Behavioral: Combined Resilience Intervention — A two-phase behavioral intervention aimed at improving psychological resilience among socioeconomically disadvantaged adolescents. The intervention includes:
  1. a 5-day structured summer camp led by trained university student volunteers, featuring psychoeducational group sessions, emotional expression activities, and life skills training, based on SEL, CBT, and positive psychology frameworks; and
  2. a 10-month pen-pal letter-writing component, where each child is matched with a trained university volunteer to receive monthly supportive letters. This stage reinforces the gains from the summer camp through sustained emotional support, skill reminders, and positive guidance.
  The intervention is designed to be low-cost, scalable, and ethically safe, and has been standardized through manuals and training protocols.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a combined intervention of summer camp and letter-writing support works to improve psychological resilience in disadvantaged adolescents in Liangshan, Sichuan. The main questions it aims to answer are:

Does the "summer camp + letter-writing" intervention improve resilience in adolescents who face poverty, lack of parental care, or social risks?

Does this intervention reduce depression and anxiety symptoms?

Researchers will compare adolescents who join the summer camp and receive monthly letters to those who do not receive this program to see if the intervention helps their mental health and coping skills.

Participants will:

Attend a 5-day summer camp that includes group games, emotion expression activities, life education, and learning support

Receive monthly letters from trained university student volunteers for about 10 months after the camp. The letters will encourage them, give advice, and help them practice what they learned in the camp

Complete surveys about their resilience, depression, and anxiety before the intervention, during it, at the end, and 6 months later

This study will also look at whether the program is cost-effective, meaning if it brings mental health benefits at a reasonable cost.

DETAILED DESCRIPTION:
This study will test a new way to help disadvantaged adolescents build psychological resilience. Psychological resilience means having the strength to handle challenges and stress in life. Many adolescents in Liangshan, Sichuan, face poverty, lack of parental care, or social risks, which increase their chances of depression, anxiety, and social withdrawal.

Researchers designed a program with two parts:

Summer camp (first month)

Participants will attend a 5-day summer camp held at a local school. University student volunteers will lead activities such as:

Team-building games to build trust and cooperation

Emotional expression through art, music, and storytelling

Life education and future planning to raise hope and self-confidence

Learning support and academic guidance The camp will provide a safe and supportive environment where adolescents can build positive relationships and learn skills to cope with difficulties.

Letter-writing support (after the camp, for 10 months)

After the summer camp, each participant will be paired with a trained university student volunteer. The volunteer will write a letter to the participant each month. Letters will:

Encourage and support the participant emotionally

Remind them to use the skills learned during the camp

Share stories, advice, and caring words to reduce loneliness

Participants will be randomly assigned to either the intervention group, who will join the camp and receive letters, or the control group, who will continue their normal school life without this program. All participants will complete surveys before the program, halfway through, at the end, and 6 months later to measure:

Psychological resilience

Depression symptoms

Anxiety symptoms

The study will also check if this program is safe, acceptable to adolescents, and cost-effective. There are no known major risks. The program does not replace professional therapy but provides social and emotional support. If any participant shows signs of severe mental health issues, the research team will help them get professional care.

This study aims to find out if combining a short-term camp with long-term letter-writing support can sustainably improve adolescents' mental health in low-resource areas. If proven effective, it may offer a scalable and low-cost way to support disadvantaged youth in rural China.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in Grade 7 or Grade 8 (junior middle school) in selected schools in Yuexi County, Liangshan Prefecture, Sichuan Province.
* Identified as "children in adversity," including those from economically disadvantaged families, left-behind children, children with disabilities, or other children deemed at-risk by school officials.
* Able to understand and complete psychological questionnaires.
* Mentally and physically able to participate in group activities and engage in written communication.
* Willing to participate in the study and provide informed assent.
* Legal guardian has signed written informed consent for participation.

Exclusion Criteria:

* Children with serious psychiatric or developmental disorders (e.g., autism spectrum disorder, intellectual disability) that impair comprehension or participation.
* Currently receiving professional psychological counseling or treatment that may interfere with the study protocol.
* Participation in other mental health interventions in the past year.
* Planning to transfer, drop out, or leave the region during the study period.
* Judged by the research team to be unsuitable for participation due to medical or other reasons (e.g., serious physical illness that prevents participation in camp activities).

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 497 (Estimated)
Dates: Start 2025-08-17 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Psychological resilience (RSCA score) at post-intervention | At baseline (1 month before intervention), mid-intervention (Month 6), end of intervention (Month 11), and follow-up (Month 17)
  Psychological resilience will be assessed using the Resilience Scale for Chinese Adolescents (RSCA), a 27-item validated instrument measuring five dimensions of resilience. Each item is rated on a 5-point Likert scale, and the total score ranges from 27 to 135, with higher scores indicating greater resilience.

SECONDARY OUTCOMES:
Change in depressive symptoms from baseline to follow-up (PHQ-9) | At baseline (1 month before intervention), mid-intervention (Month 6), end of intervention (Month 11), and follow-up (Month 17)
  Depressive symptoms will be measured using the 9-item Patient Health Questionnaire (PHQ-9), a validated screening tool for depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day), with a total score range of 0-27. Higher scores indicate more severe depressive symptoms. Clinically significant depression is defined as a score ≥10.
Change in anxiety symptoms from baseline to follow-up (GAD-7) | At baseline (1 month before intervention), mid-intervention (Month 6), end of intervention (Month 11), and follow-up (Month 17)
  Anxiety symptoms will be assessed using the 7-item Generalized Anxiety Disorder scale (GAD-7), a validated self-report measure for generalized anxiety. Each item is rated from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21. A score of ≥10 is considered clinically significant.
Change in mobile device addiction symptoms from baseline to follow-up (SAS-SV) | Baseline (T0): 1 month before summer camp Post-intervention (T2): Month 11 Follow-up (T3): Month 17
  Digital device addiction will be assessed using the Short Version of the Smartphone Addiction Scale (SAS-SV), adapted for general mobile device use. The scale includes 10 items rated on a 6-point Likert scale (1 = strongly disagree to 6 = strongly agree). Higher scores indicate greater risk of device addiction. A total score above 32 is considered indicative of problematic use.

OTHER OUTCOMES:
Change in life satisfaction from baseline to follow-up | At baseline (1 month before intervention), end of intervention (Month 11), and follow-up (Month 17)
  Life satisfaction will be assessed using a brief validated adolescent life satisfaction scale. Participants rate their overall satisfaction with life on a 5-point Likert scale. Higher scores indicate greater life satisfaction.
Change in future orientation from baseline to follow-up | At baseline (1 month before intervention), end of intervention (Month 11), and follow-up (Month 17)
  Participants' future orientation will be assessed using a brief validated scale measuring goal-setting, planning, and optimism toward future outcomes. Higher scores reflect stronger future orientation.

IPD SHARING:
Plan to Share IPD: No
This study involves vulnerable child participants, and individual-level data will not be shared due to ethical and privacy concerns. Only aggregate-level results will be made available in publications or upon request.